CLINICAL TRIAL: NCT03115398
Title: A Simple Walking Program to Enhance Concurrent Chemoradiotherapy Delivery: A Randomized Trial
Brief Title: A Simple Walking Program to Enhance Concurrent Chemoradiotherapy Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017-7472
Record Dates: First submitted 2017-03-30; First posted 2017-04-14 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Brain Cancer; Head and Neck Cancer; Lung Cancer; Gastrointestinal Cancer; Cervical Cancer
Keywords: Fitness Tracker; Activity Monitoring; Chemotherapy; Radiation Therapy; Chemoradiotherapy
MeSH Terms: conditions — Brain Neoplasms; Head and Neck Neoplasms; Lung Neoplasms; Gastrointestinal Neoplasms; Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Activity Monitoring with Routine Care (No Intervention): Subjects randomized to the control arm will wear activity trackers but will have no specific instructions to increase their activity levels.
- Pedometer-based Walking Program (Experimental): Subjects randomized to the experimental arm will be instructed to meet the customized daily step count goals that are displayed on their fitness trackers. Patients who fail to meet their step count goal for three consecutive days will be contacted by a study coordinator and reminded to try to meet the activity goals. If the patient reports that his or her activity is limited by treatment-related toxicities, the patient's treating physicians will be notified to ensure that supportive care needs are being met.
  Interventions: Behavioral: Pedometer-based Walking Program

INTERVENTIONS:
Behavioral: Pedometer-based Walking Program — Patients will be instructed to meet the daily step count goal displayed on their fitness tracker. If goal is not being met, study team will intervene and reinforce the importance of meeting this goal. Intervention will include a conversation with the patient, led by a study coordinator, to identify any challenges present in meeting the prescribed goal. Solutions to such challenges may be offered by the coordinator or necessary provider, such as a dietitian, when applicable.
  Arms: Pedometer-based Walking Program

SUMMARY:
By utilizing fitness trackers, this study aims to demonstrate that a simple walking program improves patients' ability to tolerate curative concurrent chemoradiotherapy without treatment interruption.

DETAILED DESCRIPTION:
Patients will be given a commercially available fitness tracker to wear continuously throughout the course of the study. Per this study's inclusion criteria, all patients will be treated with concurrent chemoradiotherapy for a malignancy of the brain, head and neck region, lung, gastrointestinal tract, or cervix. Patients will be randomized to one of two arms: an experimental arm, where they will be instructed to meet a daily, customized step count goal, or a control arm where they will wear activity trackers but be given no specific instructions to increase their activity levels. Patients in the experimental arm who fail to meet their step count goal for three consecutive days will be contacted by a study coordinator and reminded to try to meet the activity goals. If the patient reports that his or her activity is limited by treatment-related toxicities, the patient's treating physicians will be notified to ensure that supportive care needs are being met. With such a program, this study aims to demonstrate the potential to improve patients' ability to tolerate curative concurrent chemoradiotherapy without treatment interruption.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* ECOG performance status 0-2
* Able to ambulate independently (without the assistance of a cane or walker)
* Diagnosis of invasive malignancy of the brain, head and neck region, lung, gastrointestinal tract, or uterine cervix
* Planned treatment with fractionated (≥15 treatments) external beam radiotherapy with concurrent chemotherapy (or cetuximab) with curative intent (including preoperative or postoperative treatment)
* Women of childbearing potential must:
* Have a negative serum or urine pregnancy test within 72 hours prior to the start of study therapy
* Agree to utilize an adequate method of contraception throughout treatment and for at least 4 weeks after study therapy is completed
* Be advised of the importance of avoiding pregnancy during trial participation and the potential risks of an unintentional pregnancy.
* All patients must sign study specific informed consent prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2017-02-16 (Actual); Primary Completion 2020-03-03 (Actual); Study Completion 2021-03-03 (Actual)

PRIMARY OUTCOMES:
Number of Missed Scheduled Radiotherapy Treatments | During chemoradiotherapy (an average of 6 weeks)
  The primary endpoint of this study is missing two or more scheduled external beam radiotherapy treatments. Treatments that are cancelled due to national holidays, inclement weather, or machine issues will not count towards this endpoint.

SECONDARY OUTCOMES:
Daily Step Counts | During chemoradiotherapy and over the following 4 weeks (an average of 10 weeks)
  Step counts will be recorded and measured daily from patients' fitness trackers.
Treatment-related Toxicities | During chemoradiotherapy and over the following 4 weeks (an average of 10 weeks)
  Toxicities will be evaluated each week and scored using CTCAE version 4.03.
Patient-reported Quality of Life Scores | During chemoradiotherapy and over the following 4 weeks (an average of 10 weeks)
  Measured weekly using the EORTC QLC-C30.
Number of Emergency Room Visits | During chemoradiotherapy and over the following 4 weeks (an average of 10 weeks)
  Using the EMR, a record will be kept indicating the number of times each patient visits the emergency room.
Number of Hospitalizations | During chemoradiotherapy and over the following 4 weeks (an average of 10 weeks)
  Using the EMR, a record will be kept indicating the number of times each patient is hospitalized.
Modified Glasgow Prognostic Scores | During chemoradiotherapy and over the following 4 weeks (an average of 10 weeks)
  Scores will be calculated based on serum albumin and C-reactive protein levels.
Disease Progression or Recurrence | Through study completion, an average of 1 year
  Disease progression or recurrence, to be scored by treating physicians based on available clinical and imaging data
Survival Status | Through study completion, an average of 1 year
  Survival data will be kept for all patients on study throughout treatment and follow-ups.

CONTACTS AND LOCATIONS:
Overall Officials: Nitin Ohri, MD, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No